CLINICAL TRIAL: NCT06641921
Title: A Multi-centre, Prospective, Single-arm, Open-label Trial With a Prespecified Effectiveness Endpoint to Evaluate the Benefits of Haemodynamically Guided Treatment Using the Seerlinq HeartCore System in Heart-failure Patients.
Brief Title: Strategy TO Prevent Decompensated Heart Failure
Acronym: #STOP-DHF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seerlinq s. r. o. (Other)
Collaborators: Premedix Academy (Other); Premedix Clinic (Unknown); Dôvera zdravotná poisťovňa, a.s. (Unknown); LA-RO COR (Unknown); KardioNitra Ambulancia (Unknown); Nemocnica s poliklinikou, Nové Mesto nad Váhom, n. o. (Unknown); Kardiologia KK (Unknown); Interná a kardiologická ambulancia Trebišov, spol. s r.o. (Unknown); Nemocnica Hlohovec (Unknown); KCNR (Unknown); Kardiocomp (Unknown); Mydliar Intermedical (Unknown); Súscch (Unknown); NAW - Nemocnica Piestany (Unknown); IMCORE, s.r.o (Unknown); Diagnos - SM, s.r.o. (Unknown); Interna a diabetologicka ambulancia Skalica (Unknown); UPJS Kosice (Unknown); BalMedic s.r.o. (Unknown); SUSCCH (Unknown); KCNR - Trnava / Nemocnica NMnV (Unknown); FN Trenčín (Unknown); K+R (Unknown); DevinAmb / Kardio-Sanus (Unknown); UNB Ruzinov (Unknown); Nemocnica s poliklinikou v Rožňave - Penta Hospitals (Unknown); NemoSan (Unknown); Duo Medical sro (Unknown); Valys s.r.o. (Unknown); CARDIOCONSULT s.r.o. (Unknown); Sciens s.r.o. (Unknown); NsP Bardejov (Unknown); KCNR, Kardiologická ambulancia, Trnava (Unknown); FNsP J. A. Reimana Prešov (Unknown); NUSCH (Unknown); FN Nitra (Unknown); Poliklinika Karlova Ves (Unknown); Nemocnica s Poliklinikou Čadca (Unknown); Nemocnica Staré mesto - UNB - Mickiewiczova (Unknown); Nemocnica Poprad (Unknown); Semper Cor s.r.o. (Unknown); Nemocnica Milosrdni Bratia (Unknown); MediKardio (Unknown); CorDei (Unknown); NNG Bory (Unknown); Nemocnica Považská Bystrica (Unknown); NsP Sv. Jakuba, n.o., Bardejov (Unknown); Ščasná, s.r.o. (Unknown); NSP Myjava (Unknown); Nemocnica Partizánske (Unknown); Dom srdca s.r.o. (Unknown); Nemocnica s poliklinikou Dunajská Streda, a.s. (Unknown); CorArt s.r.o. (Unknown); Nemocnica Malacky (Unknown); Solikcardiology (Unknown); Samaria (Unknown); NspBr (Unknown); East Slovak Institute for Cardiovascular Diseases (Other); KARDIOPREVENT (Unknown); Sabimed (Unknown); Fakultná nemocnica s poliklinikou Nové Zámky (Unknown); Sukr Amb v Ružinovskej poliklinike - MUDr O.B. s.r.o. (Unknown); Barmeda (Unknown); MD clinic (Unknown); Marmedico (Unknown); Nemocnica s poliklinikou Spišská Nová Ves a.s. (Unknown); M.K.U. Med (Unknown); AJC MED, s.r.o. (Unknown); Luxicor s.r.o. (Unknown); Interna Zvolen s.r.o. (Unknown); ŽILPO (Unknown); INTER - KARDIO, s.r.o. (Unknown); KVC - Kardiovaskulárne Centrum s.r.o. (Unknown); Hospitale s.r.o. (Unknown); Klinika Orbis (Unknown); FNsP BB (Unknown); Polymedica - Praha (Unknown); Neštátna interná ambulancia - MUDr. O.K. (Unknown); Poliklinika ŽnH (Unknown); Veria s.r.o. (Unknown); UNM - Univerzitná nemocnica Martin (Unknown); Delio spol. s.r.o. (Unknown); Ortovita (Unknown); CINRE (Unknown); Kardiologická ambulancia, MUDr. MG, Michalovce (Unknown); Nemocnica Skalica (Unknown); Operatíva, lekárska spoločnosť, spol. s r.o. (Unknown); P&P MEDINE s.r.o. (Unknown); Zdravie Martin s.r.o. (Unknown); CARDIO s.r.o. (Unknown); Kardio-Sanus (Unknown); Kardio ZM (Unknown); OMCOR s. r. o. (Unknown); Kardio R s.r.o. (Unknown); ZK Cardio ambulancia (Unknown); UN Martin (Unknown); REKA Kežmarok, s.r.o. (Unknown); JM Interna (Unknown); IV. interná klinika LF UK a UNB (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 012024
Record Dates: First submitted 2024-10-08; First posted 2024-10-15 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure; Remote Monitoring
Keywords: heart failure; remote monitoring; photoplethysmography; telemedicine
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Seerlinq intervention arm (Experimental): Participants in the intervention arm will be haemodynamically-guided based on the results from the Seerlinq telemedical monitoring system.
  Interventions: Device: Seerlinq Telemedical Monitoring System

INTERVENTIONS:
Device: Seerlinq Telemedical Monitoring System — Participants will use the Seerlinq telemedical monitoring system and receive standardized remote training to perform regular photoplethysmography (PPG) measurements and symptom reporting. Heart failure management will be hemodynamically guided, with treatment decisions based primarily on trends in estimated left ventricular filling pressure (LVFP) derived from Seerlinq. The therapeutic goal is to reduce elevated LVFP through adjustment of diuretics, vasodilators, or neurohormonal agents. Additional parameters-including heart rate, patientreported fatigue and shortness of breath, and home blood pressure values-will support individualized therapy titration. If elevated LVFP persists despite remote treatment adjustments, patients will be scheduled for inperson clinical evaluation. Guidelinedirected medical therapy (GDMT) will be uptitrated according to hemodynamic tolerance following a prespecified treatment protocol aligned with current heart failure management guidelines. .

SUMMARY:
The goal of this prospective, multicenter, single-arm, open-label clinical trial (Strategy TO Prevent Decompensated Heart Failure) is to evaluate the 6month incidence of heart failure hospitalization (HFH) and all cause mortality in patients managed with haemodynamically guided treatment using the Seerlinq telemedical monitoring system.

DETAILED DESCRIPTION:
Study participants will receive the Seerlinq telemedical monitoring system with appropriate training and will perform regular measurements as instructed. HF treatment will be haemodynamically-guided, with clinical decisions informed by trends in LVFP determined by Seerlinq. The primary treatment goal will be to lower elevated LVFP using diuretics, vasodilators, or neurohormonal agents. In addition to LVFP, treatment decisions will be supported by heart rate, patient perceived symptoms (fatigue and shortness of breath) and blood pressure values measured using a certified home blood pressure monitor, enabling more individualized titration of therapy based on a comprehensive haemodynamic profile. In cases where elevated LVFP persists despite treatment adjustments and consultation with a healthcare professional via telephone, or where there is evidence of non-response, patients will be promptly scheduled for an urgent in-person clinical evaluation to assess fluid status, comorbidities, and potential treatment barriers. Furthermore, the Seerlinq-guided approach will aim for the accelerated uptitration of guideline-directed medical therapy (GDMT) based on haemodynamic tolerance. Haemodynamically guided management will be conducted according to a prespecified protocol (Treatment Protocol) in line with current guidelines for management of chronic heart failure

ELIGIBILITY:
Inclusion Criteria

1. Males and females aged ≥ 18 years.
2. Able to understand, and willing to provide written informed consent.
3. Stated willingness to comply with all study procedures and lifestyle considerations and availability for the duration of the study.
4. Diagnosis of chronic heart failure in NYHA class II or III
5. Able to stand for 2 minutes
6. Access to necessary resources for participating in a technology-based intervention (smartphone, blood pressure monitor, internet access).

Exclusion Criteria

The participant may not enter the study if ANY of the following apply:

1. Use of other services for telemedical monitoring for heart failure.
2. Renal failure with a Glomerular Filtration Rate (GFR) <25 ml/min or requiring renal replacement therapy.
3. Pregnancy, female participant lactating or planning pregnancy during the course of the trial.
4. Complex congenital heart disease
5. Subjects with known pulmonary hypertension (WHO category 1 or 3/4/5)
6. Inability to perform regular measurements alone or with help of a caregiver.
7. Other possible unforeseen medical conditions that the investigator deems unsafe for study participation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
Heart failure hospitalization and mortality | in 6 months
  Composite incidence of heart-failure hospitalization or all-cause mortality during an average follow-up of 6 months, assessed against a prespecified performance goal (PG) of 9.0 %

SECONDARY OUTCOMES:
Number of hospitalizations for HF | in 6 months
  Rate of heart failure hospitalization in 6 month
Medication changes | in 6 months
  Any medication changes triggered by remote monitoring
Telephone contacts | in 6 months
  Total count of medical telephone contacts documented between investigational sites and participating patients triggered by remote monitoring.
Cardiology visits | in 6 months
  Total number of in-person cardiology visits triggered by monitoring
Patient compliance | in 6 month
  Patient compliance with device measurement.

OTHER OUTCOMES:
Health care costs | in 6 month
  Total healthcare costs per patient associated with management during the average 6-month follow-up period.
Incremental cost-effectiveness ratio | in 6 months
  Incremental cost-effectiveness ratio (ICER): cost per avoided heart-failure hospitalization or all-cause mortality event at 6 months.
Healthcare resource-utilization costs | in 6 months
  Healthcare resource-utilization costs per patient, including expenditures for heart-failure hospitalizations, emergency-department visits, outpatient consultations, and medication adjustments over the follow-up period
Comparison of healthcare costs between Seerlinq-guided management and standard-of-care | in 6 month
  Comparison of total healthcare costs per patient between Seerlinq-guided management and the propensity score-matched standard-of-care (SOC) cohort over the same follow-up duration.

CONTACTS AND LOCATIONS:
Overall Officials: Allan Böhm, MD, Principal Investigator — Seerlinq
Locations (1):
- Premedix Clinic, Bratislava, Nové Mesto, Slovakia

IPD SHARING:
Plan to Share IPD: Undecided